CLINICAL TRIAL: NCT07243379
Title: A Prospective Real-World Observational Study of Nanocrystalline Megestrol Acetate in Patients With Cancer Cachexia
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Changchun GeneScience Pharmaceutical Co., Ltd. (Industry)
Collaborators: Henan Cancer Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Megaxia-RWS 01
Record Dates: First submitted 2025-11-15; First posted 2025-11-21 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-10

CONDITIONS: Clinical Characteristics and Treatment Outcomes of Malignant Tumor Cachexia; Multicenter Observational Study

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Nanocrystalline Megestrol Acetate Oral Suspension + Standard Antitumor Therapy (Experimental): This cohort focuses on patients who have already been diagnosed with cachexia before the initiation of this study and are scheduled to receive treatment with nanocrystalline megestrol acetate.
  Interventions: Drug: Nanocrystalline Megestrol Acetate

INTERVENTIONS:
Drug: Nanocrystalline Megestrol Acetate — Nanocrystalline Megestrol Acetate oral suspension, with a specification of 125 mg/mL, administered orally at a dose of 5 mL per day (625 mg/day), and the primary endpoint efficacy collection will be conducted in the 4th week.

SUMMARY:
This study is a prospective, real-world observational study. The objective is to evaluate the effectiveness and safety of nanocrystalline megestrol acetate in patients with cancer cachexia in real-world settings. Eligible participants were patients diagnosed with cancer cachexia who were scheduled to receive treatment with nanocrystalline megestrol acetate.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically and/or cytologically confirmed malignancy.
* Age ≥18 years at enrollment.
* Eastern Cooperative Oncology Group (ECOG) performance status score of 0-2 and an expected survival of ≥3 months.
* Meeting the diagnostic criteria for cachexia (based on Fearon's criteria).
* Body mass index (BMI) ≤30.

Exclusion Criteria:

* Presence of any condition affecting gastrointestinal absorption, such as dysphagia, malabsorption, or uncontrolled vomiting; patients receiving tube feeding or parenteral nutrition.
* Presence of anorexia due to anorexia nervosa, psychiatric disorders, or pain that makes eating difficult.
* Patients with acquired immunodeficiency syndrome (AIDS).
* Currently receiving or planning to receive other medications that increase appetite or body weight, such as corticosteroids (except short-term dexamethasone during chemotherapy), androgens, progestins, thalidomide, olanzapine, anamorelin, or other appetite stimulants.
* Patients with Cushing's syndrome, adrenal or pituitary insufficiency, or poorly controlled diabetes mellitus.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 495 (Estimated)
Dates: Start 2025-09-25 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with improved appetite at Week 4 based on the A/CS-12 scale. | Week 4

SECONDARY OUTCOMES:
Proportion of patients with >5% increase in body weight from baseline at Week 4, Week 8, and Week 12. | Proportion of patients with >5% increase in body weight from baseline to week 12.

CONTACTS AND LOCATIONS:
Locations (1):
- Henan Cancer Hospital, Affiliated to Zhengzhou University, Zhengzhou, Henan, China